CLINICAL TRIAL: NCT02405429
Title: Comparing Temporal Artery and Axillary Temperatures With Rectal Temperature in Neonates
Brief Title: Temporal Artery Temperature Measurement in Neonates
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Edward F. Bell, Professor of Pediatrics, University of Iowa
Other Study IDs: 201404832
Record Dates: First submitted 2015-03-25; First posted 2015-04-01 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Newborn Infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to evaluate the temporal artery thermometer by comparing temporal artery and axillary thermometer temperature measurements with rectal thermometer temperature measurements in neonatal patients. The investigators measured temporal artery, axillary, and rectal temperatures of 49 infants. Temporal artery temperature was measured using an infrared temporal artery thermometer, and the results with this device were compared with axillary temperature (clinical standard) and rectal temperature (gold standard). The difference between rectal and temporal artery temperatures was compared with the difference between rectal and axillary temperatures for each infant, and the data were analyzed based on weight, postmenstrual age and bed type - open crib or incubator.

ELIGIBILITY:
Inclusion Criteria:

* Patients in hospital well-baby nursery or neonatal intensive care unit

Exclusion Criteria:

* Birth weight <500 grams
* Anal atresia
* Central nervous system malformation
* Hypoxic-ischemic encephalopathy
* Clinical concerns for necrotizing enterocolitis or other bowel injury or discontinuity

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Hospital nursery patients
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Bell, MD, Principal Investigator — University of Iowa

REFERENCES:
- [Result] Syrkin-Nikolau ME, Johnson KJ, Colaizy TT, Schrock R, Bell EF. Temporal Artery Temperature Measurement in the Neonate. Am J Perinatol. 2017 Aug;34(10):1026-1031. doi: 10.1055/s-0037-1601440. Epub 2017 Apr 10. PMID 28395367

RESULTS

PARTICIPANT FLOW:
Groups:
- Hospitalized Neonates: Patients in the neonatal intensive care unit or the newborn nursery
Period: Overall Study
Arm/Group | Hospitalized Neonates
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hospitalized Neonates
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: days] | 11 [1 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 49
Gestational Age [Median (Full Range); unit: weeks] | 34 [25 to 40]
Body Weight at Time of Study [Median (Full Range); unit: grams] | 2235 [1160 to 4205]

OUTCOME MEASURES:

1. Primary Outcome: Temporal Artery Temperature
Description: With commercial infrared temporal artery thermometer
Time Frame: Mean of 2 measurements within 2 minutes of each other and within 2 minutes of axillary and rectal temperature measurements
Population: Hospitalized neonates
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Hospitalized Neonates
Number analyzed (Participants) | 49
degrees Celsius | 37.16 (0.36)

2. Primary Outcome: Axillary Temperature
Description: With commercial digital thermometer
Time Frame: Single measurement within 2 minutes of temporal artery and rectal temperature measurements
Population: Hospitalized neonates
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Hospitalized Neonates
Number analyzed (Participants) | 49
degrees Celsius | 36.61 (0.30)

3. Primary Outcome: Rectal Temperature
Description: With thermistor probe and telethermometer
Time Frame: Single measurement within 2 minutes of temporal artery and axillary temperature measurements
Population: Hospitalized neonates
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Hospitalized Neonates
Number analyzed (Participants) | 49
degrees Celsius | 36.82 (0.30)

4. Primary Outcome: Difference Between Temporal Artery and Rectal Temperatures
Description: Rectal temperature minus temporal artery temperature
Time Frame: Within 2 minutes of each other
Population: Hospitalized neonates
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Hospitalized Neonates
Number analyzed (Participants) | 49
degrees Celsius | -0.34 (0.37)

5. Primary Outcome: Difference Between Rectal and Axillary Temperatures
Description: Rectal temperature minus axillary temperature
Time Frame: Within 2 minutes of each other
Population: Hospitalized neonates
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Hospitalized Neonates
Number analyzed (Participants) | 49
degrees Celsius | 0.21 (0.26)

ADVERSE EVENTS:
Arm/Group | Hospitalized Neonates
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No